CLINICAL TRIAL: NCT01715974
Title: Administration of GM-CSF in Women With Recurrent Implantation Failure in IVF Cycles and Egg Donation Cycles
Brief Title: Use of GM-CSF Treatment in Recurrent Implantation Failure
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre for Endocrinology and Reproductive Medicine, Italy (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HC0003
Record Dates: First submitted 2012-03-02; First posted 2012-10-29 (Estimated); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Women With Recurrent Implantation Failure in IVF
Keywords: GM-CSF, IVF failure,pregnancy
MeSH Terms: interventions — Granulocyte-Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CONTROL (Placebo Comparator): patients with recurrent implantation failure treated with PLACEBO (saline solution) from the day of embryo transfer through the day of beta hCG test
  Interventions: Drug: CONTROL
- GM-CSF group (Experimental): patients with recurrent implantation failure treated with GM-CSF (30 micrograms/day) from the day of embryo transfer through the day of beta hCG test
  Interventions: Drug: GM-CSF group

INTERVENTIONS:
Drug: GM-CSF group — 30 micrograms/day of GM-CSF from the day of embryo transfer through the day of beta HCG test
  Other Names: GM-CSF
  Arms: GM-CSF group
Drug: CONTROL — saline infusion every day from the day of embryo transfer through the day of beta HCG test
  Other Names: SALINE INFUSION
  Arms: CONTROL

SUMMARY:
The purpose of this study is to determine whether in Assisted Reproductive Technologies the treatment with GM-CSF, a growth factor working on stem cells, may improve the pregnancy rate and pregnancy outcome in patients experiencing recurrent implantation failure in IVF cycles.

DETAILED DESCRIPTION:
The GM-CSF is a cytokine promoting leukocyte growth, but also trophoblast development. In this randomized sudy investigators will test this cytokine as a treatment for recurrent implantation failure after IVF, at leat three failed previous IVF attempts.

The study will be conducted in 100 women with recurrent implantation failure of egg donation cycles. The inclusion criteria will be, at least three previous failed Egg Donation attempts where at least 4 good blastocysts were transferred, women less than 50 years old, absence of systemic diseases. These women will undergo egg donation cycle and they will randomly divided in two groups: one (50 women) will be treated with subcutaneous GM-CSF 60 micrograms/day from the day of transfer to the day of β-hCG test, and if it will be positive the treatment will be continued for other 40 days; the group of control will be treated with subcutaneous saline solution infusion in the same way of the study group. Primary outcomes will be considered: pregnancy rate and live birth rate, the of β-hCG levels at 14/21/28 and 35 days after embryo transfer.

ELIGIBILITY:
Inclusion Criteria:

* women 50 years old or less with three or more previous egg donation cycles failed,
* with a total of at least 4 blastocysts replaced in uterus

Exclusion Criteria:

* chromosomal defects in the patients,
* metabolic diseases (diabetes etc.)
* genetic diseases (thalassemia, cystic fibrosis, etc.)

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2017-12-12 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
pregnancy outcome | 12 months
  The number of patients pregnant after treatment with GM-CSF (30 microgram/day)compared with the number of patients pregnant in the control group

SECONDARY OUTCOMES:
implantation rate | 12 months
  number of embryos implanted

CONTACTS AND LOCATIONS:
Overall Officials: Marco Sbracia, MD, Study Chair — Centre for Endocrinology and Reproductive Medicine, Italy
Locations (1):
- Cerm-Hungaria, Rome, Italy

REFERENCES:
- [Background] Scarpellini F, Sbracia M. Use of granulocyte colony-stimulating factor for the treatment of unexplained recurrent miscarriage: a randomised controlled trial. Hum Reprod. 2009 Nov;24(11):2703-8. doi: 10.1093/humrep/dep240. Epub 2009 Jul 17. PMID 19617208
- [Derived] Scarpellini F, Sbracia M, Marconi D, Fracassi A, Santi K, Desole E. A Randomised Controlled Trial on the Treatment of Recurrent Implantation Failure Women Who Failed Egg Donation Cycles Using Low-Dose GM-CSF. Am J Reprod Immunol. 2025 Sep;94(3):e70162. doi: 10.1111/aji.70162. PMID 40965804